CLINICAL TRIAL: NCT04087590
Title: Impact of Inhaled PT003 on Complexity and Variability of Tidal Breathing and Oscillatory Mechanics in Stable COPD Patient
Acronym: OSCIVARI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018_24; 2018-003061-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-07-10; First posted 2019-09-12 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Copd
Keywords: long acting bronchodilator; tidal breathing; variability; impulse oscillometry spirometry; plethysmography; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PT003 treatment (Experimental)
  Interventions: Drug: Formoterol-glycopyrronium co suspension (PT003)

INTERVENTIONS:
Drug: Formoterol-glycopyrronium co suspension (PT003) — Formoterol-glycopyrronium co suspension (PT003) in a Metered Dose Inhaler, 2 puffs twice daily

SUMMARY:
Prospective, single-arm, open label, multicentre, phase II pilot study to evaluate the immediate and short term (one month) impact of a new long acting double bronchodilator on innovative parameters in stable and moderate to severe COPD patients.

* Variability and complexity of resting tidal breathing
* Oscillatory resistance and reactance of airways Tidal volume variability and complexity is decreased in airway obstruction and is expected to improve with a bronchodilator treatment, together with lung mechanics.

The relationship with changes in dyspnea and conventional pulmonary function tests is the second aim of study.

After baseline assessment of these parameters, clinical and lung function evaluation will be performed 2 hours post-drug (peak drug effects). Patients will continue treatment with PT003 for 4 weeks. On Day 30, the same clinical and lung function assessments will be performed pre (trough) and 2h-post dose in order to obtain after-treatment measurements.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 40-75 years Documented COPD in stable condition FEV1 between 30 % and 70 % predicted (post bronchodilator) Significant dyspnea with a mMRC dyspnea scale

Exclusion Criteria:

* History or current diagnosis of asthma or ACO (asthma-COPD overlap syndrome)
* Respiratory infection or COPD exacerbation within 6 weeks (2 months if it resulted in hospitalization) prior to screening
* Clinically significant or relevant cardiovascular conditions, laboratory tests, electrocardiogram (ECG) parameters
* Severe renal impairment eGFR < 30
* Narrow-angle glaucoma that, in the opinion of the Investigator, has not been adequately treated.
* Symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that is clinically significant

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Analysis of tidal volume (VT) complexity (noise limit as main parameter ) | at 1 month
  Comparison of the noise limit between V2 baseline (pre-treatment) and V3 peak (2 hours +/- 30 min post dose).
  Noise limit is a mathematical treatment of tidal breathing signal evaluating its complexity and no other description can be provided

SECONDARY OUTCOMES:
change of frequency-tidal volume pattern | Baseline, at 1 month
  the inspiratory time (Ti, measured in second) , the expiratory time (Te,measured in second) and the respiratory frequency
Tidal volume Largest Lyapunov component (an indicator of the sensitivity of the system to initial conditions) | Baseline, at 1 month
change of resistance at 5Hz , at 20 Hz | Baseline, at 1 month
  The fundamental principle of forced oscillometry is that lung function can be assessed by measuring changes in pressure and flow in response to external pressure applied at the airway opening. Resistance is complex measure that incorporates the lack of changes in pressure and volume and the rate of these changes in response to pressure oscillations at a specific frequency.
  All these measurements are expressed in the same unit (for resistance and reactance) and refer to oscillatory mechanics obtained by the same device. AX and resonant frequency are correlated to reactance.
Change of reactance | Baseline, at 1 month
  the fundamental principle of forced oscillometry is that lung function can be assessed by measuring changes in pressure and flow in response to external pressure applied at the airway opening. Reactance is complex measure that incorporates the changes in pressure and volume and the rate of these changes in response to pressure oscillations at a specific frequency at 5Hz was used. Reactance is thought to reflect the elastic properties of the lung.
  All these measurements are expressed in the same unit (for resistance and reactance) and refer to oscillatory mechanics obtained by the same device.
Change of AX and resonant frequency | Baseline, at 1 month
  Area under reactance curve (AX) and resonant frequency are correlated to reactance.
change of spirometry parameters | at 1 month
  Spirometry : FEV1, FVC, FEV1/FVC
change in lung function as assessed through body plethysmography | Baseline, at 1 month
  Change from baseline to end of treatment in the following measures Total lung capacity (TLC) Residual volume (RV) Inspiratory capacity (IC) Functional residual capacity (FRC) All plethysmographic parameters shown here are lung volumes, expressed in liters, and are somewhat interrelated. For instance IC is TLC- FRC.There is no reason to separate these outcome measures
change of airway resistance (RAW) and specific airway conductance (sGAW). | Baseline, at 1 month
  sGaw is specific conductance, ie 1/resistance divided by the volume at which resistance was measured. These two parameters are always measured and used together.
  All plethysmographic parameters shown here are lung volumes, expressed in liters, and are somewhat interrelated.
Visual Analogic Scale | Baseline, at 1 month
  Two VAS (± 100 mm ) will be used to evaluate changes (much worse-unchanged-much better) in dyspnea and chest tightness 2 hours after PT003 administration and at 4 weeks in through and post dose conditions
Likert scales | Baseline, at 1 month
  Likert scales (7 points) will assess changes in dyspnea and global health at visit 3 in comparison with pre treatment condition (V2).
BDI/TDI | Baseline, at 1 month
  The BDI/TDI is an instrument developed to provide a multidimensional measure of dyspnea in relation to activities of daily living. The Baseline Dyspnea Index (BDI) provides a measure of dyspnea at a single state, the baseline, and the Transitional Dyspnea Index (TDI) evaluates changes in dyspnea from the baseline state. The instrument consists of three components: functional impairment, magnitude of task, and magnitude of effort. For the BDI, each of these three components are rated in five grades from 0 (severe) to 4 (unimpaired), and are summed to form a baseline total score from 0 to 12. For the TDI, changes in dyspnea are rated for each component by seven grades from -3 (major deterioration) to +3 (major improvement), and are added to form a total TDI score from -9 to +9. Positive scores indicate an improvement, and a change from the BDI or a difference between treatments of 1 point has been estimated to constitute the minimum clinically important difference (MC
mMRC dyspnea scale | Baseline, at 1 month
  The Modified Medical Research Council (mMRC) dyspnea scale uses a simple grading system to assess a subject's level of dyspnea that consists of five statements about perceived breathlessness. It is an interviewer-administered ordinal scale on which subjects provide their dyspnea according to five grades of increasing severity (scores ranges from 0 (none) to 4 (very severe).
Modified Dyspnea Profile (MDP) | Baseline, at 1 month
  The MDP consists of 11 items evaluating both the sensory and affective dimensions of dyspnoea. One item (A1) assesses the unpleasantness of dyspnoea on a 0-10 visual numerical scale anchored by "neutral" (0) and "unbearable" (10). Five items assess the sensory dimension of dyspnoea, both in terms of quality and intensity (on a scale of 0-10). Five items assess the affective dimension of dyspnoea, also in terms of quality and intensity (on a scale of 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PEREZ, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Calmette Chu Lille, Lille, France